CLINICAL TRIAL: NCT05186038
Title: Scrutiny Based in a Novel Test to Help the Early Detection of Celiac Disease.
Brief Title: Mass Screening for the Early Detection of Patients With Celiac Disease.
Status: Completed | Type: Observational
Sponsor: Biomedal S.L. (Other)
Collaborators: University of Seville (Other); FUNDACION IHP (Unknown)
Responsible Party: Sponsor
Other Study IDs: CELISIN
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Celiac Disease
Keywords: Mass screening; Diagnosis; Celiac disease; Urine samples; Blood samples
MeSH Terms: conditions — Celiac Disease; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population of children and adolescents between 2 and 18 years old: Population of children and adolescents between 2 and 18 years old who are diagnosed with celiac disease or are suspected to suffer the disease.
  Interventions: Diagnostic Test: iVYCHECK GIP Urine; Diagnostic Test: CeliacDetect

INTERVENTIONS:
Diagnostic Test: iVYCHECK GIP Urine — To determine the presence of Gluten Immunogenic Peptides (GIP) in urine samples using the immunochromatographic test iVYCHECK GIP Urine (Biomedal S.L).
Diagnostic Test: CeliacDetect — To determine the presence of IgA anti-tTG antibodies in blood samples using the immunochromatographic test CeliacDetect (Biomedal S.L).

SUMMARY:
The use of a home rapid test for the detection of both gluten immunogenic peptides (GIP) in urine and immunoglobulin A (IgA) anti tissue transglutaminase (anti-tTG) antibodies in blood may contribute to the early detection of volunteers who suffer celiac disease (CD), a highly under-diagnosed disorder. Patients with positive results could inform their doctors in order to accelerate the diagnosis, contribute to symptoms control and improve their quality of life.

This observational, cross-sectional study with no interventions applied in subjects consists on a single group of volunteers between 2 and 18 years old. They will be given an informed consent which must be signed by them or their parents/legal guardians, a Celiac Symptoms Index (CSI) questionnaire and the sample collection material required on the testing day. Urine samples will be collected and analysed in situ or alternatively they will be stored and analyzed after at the laboratory. Blood samples will be collected and analyzed in situ the testing day.

The main outcome is to determine the prevalence of CD through mass screening within the pediatric and adolescent population in order to provide an early diagnosis and avoid long-term consequences which are suffered by untreated patients. As an international innovation, misdiagnosis (false negatives) because of an insufficient gluten intake are expected to be detected, thus the use of GIP detection in urine will confirm gluten ingestion at the diagnosis. Volunteers with a confirmed diagnosis of CD could be monitored by their doctors to corroborate whether a gluten-free diet improves their quality of life.

DETAILED DESCRIPTION:
Hypothesis: the use of a home rapid test for the detection of both gluten immunogenic peptides (GIP) in urine and IgA anti-tTG antibodies in blood may contribute to the early detection of volunteers who suffer celiac disease (CD), a highly under-diagnosed disorder. Patients with positive results could inform their doctors in order to accelerate the diagnosis, contribute to symptoms control and improve their quality of life.

Objectives:

Primary objective: to perform a mass screening in the pediatric and adolescent population (2 - 18 years old) in order to assess the prevalence of the CD providing early diagnosis of possible patients through 1 - Detection of IgA anti-tTG antibodies present in blood (to be measured by home rapid tests); 2 - Detection of GIP in urine (to be measured in situ or at a central laboratory).

Specific objectives: 1- To determine the prevalence of CD, particularly in children between 2 and 18 years old; 2 - To detect possible hidden CD cases, avoiding future irreversible damages by a late detection of this pathology such as growth impairment, decalcification, neurotoxicity or risks of suffering other autoimmune diseases; 3 - To detect misdiagnosis (false negatives) because of an insufficient gluten intake, as an international innovation.

Study design: this observational, cross-sectional study with no interventions applied in subjects consists of a single group of volunteers between 2 and 18 years old. They will be given an informed consent which must be signed by them or their parents/legal guardians, a Celiac Symptoms Index (CSI) questionnaire, a short clinical questionnaire and the sample collection material required on the testing day. Urine samples will be collected and analysed in situ or alternatively they will be stored and analyzed after at the laboratory. Blood samples will be collected and analyzed in situ the testing day.

Study participants: volunteers from the pediatric and adolescent population between 2 and 18 years old. Gluten consumption previous to testing is an innovative requirement in order to validate the IgA anti-tTG antibodies rapid test.

Study procedure:

1. Patient enrollment.
2. Testing day: all participants will 1 - return the informed consent signed by them or their parents/legal guardians; 2 - complete the Celiac Symptoms Index (CSI) questionnaire and the clinical questionnaire to check if they have had any previous symptoms or other relevant information to be considered; 3 - collect urine samples in order to determine GIP presence through a immunochromatographic test (iVYCHECK GIP Urine, Biomedal S.L., Seville, Spain) in situ or at the central laboratory, therefore samples will need to be stored. It may be confirmed whether the volunteer was ingesting gluten when the test was performed. - A. If the result is positive, a serological test will be performed at a certified laboratory in order to confirm the volunteer's disease and a specialist to perform the diagnosis will be recommended. Whether the diagnostic is confirmed, five GlutenDetect's units will be given to each diagnosed volunteer to make sure they can check whether the diet is properly followed. - B. If the result is negative, the possibilities of suffering CD are low so any additional test will be performed. Exceptionally, those whose gluten level in urine is undetectable, but their CeliacDetect result appears as negative, a deeper study will be performed about gluten ingestion the day before through 24 hours recall.

Number of participants: a minimum of 1000 volunteers would be needed to achieve a conclusive study in order to determine at least 10 cases of CD. The calculation was made according to CD's prevalence of 1% described by several studies.

Measurements: 1- Laboratory rapid test (iVYCHECK GIP Urine, Biomedal S.L., Seville, Spain) for GIP determination in urine samples and immunochromatographic rapid test (CeliacDetect, Biomedal S.L., Spain) for IgA anti-tTG antibodies detection in blood; 2- CD related symptoms (CSI questionnaire). Urine samples will be analysed in situ or stored and analyzed later at a central laboratory (Biomedal S.L., Seville, Spain).

Statistical analysis: the data obtained in the study will be collected in a data base created with this purpose. Variables are tabulated through the IBM SPSS Statistics V25.0 program from International Business Machines (IBM) (Armonk, New York, USA). Different study variables will be considered: 1 - related to patients (age, gender, parent's study level); 2 - related to the "Celiac symptoms index" questionnaire (presence or not of previous symptomatology); 3 - related to samples (GIP presence in urine and IgA anti-tTG antibodies presence in blood). Each test's result will be considered as significant if the value p<0,05 and very significant if p<0,01. A confidence of 95% will be taken for intervals. When p>0,05, the result will be considered as non-significant.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents volunteers (2-18 years old).
* Regular gluten consumption.
* Willingness to perform the study and ability to collect urine samples.
* The signing of the informed consent by the volunteer and his/her legal guardians.

Exclusion Criteria:

* Related diseases or psychiatric alterations which do not recommend being included in the study as the researcher's consideration.
* Lack of foreseeable collaboration.
* Patients which do not provide samples or surveys in 70% of cases.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Population comprised of patients between 2 and 18 years old who are diagnosed with celiac disease or suspected to suffer the disease. They should have willingness to perform the study and ability to collect urine samples. Moreover, the patients or their legal guardians have to sign the informed consent.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-12-18 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Presence of Gluten Immunogenic Peptide (GIP) in urine | Only the testing day.
  The immunochromatographic test iVYCHECK GIP Urine allows the detection of GIP resulting from gastrointestinal degradation of ingested gluten in urine. The detection step is based on the reaction of the 33-mer-like immunogenic peptides of gluten present in the sample with the coloured conjugated (monoclonal anti-gliadin 33-mer antibody/red-coloured microsphere) previously loaded in the cassette. Complexes spread through the cassette by capillarity and interact with a second anti-gliadin 33-mer antibody immobilized on the membrane at the test zone. A red line at the test zone indicates a positive result while the absence of the red line indicates a negative result.
Presence of IgA anti-tTG in blood | Only the testing day.
  The immunochromatographic test CeliacDetect allows the detection of IgA anti-tTG in blood samples. The detection step is based on the union of the IgA anti-tTG with anti human IgA antibodies labeled with colloidal gold and tTG (whose origin is the erythrocyte lysis in the dilution buffer). The complex would be bounded to the stable protein line (test line) by tTG. A red line at the test zone indicates a positive result while the absence of the red line indicates a negative result.

SECONDARY OUTCOMES:
Presence of previous symptoms | Only the testing day.
  Number of participants with CD symptoms previously to the study as assessed by Celiac Symptoms Index (CSI) questionnaire. The scores on the CSI are recoded into a scale from 16 to 80. A score of ≥38 is considered as symptomatic.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Salamanca, Study Chair — FUNDACION IHP
Locations (2):
- Spain (2):
  - 37th Celiac Festival, Madrid
  - Grupo IHP, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Husby S, Koletzko S, Korponay-Szabo IR, Mearin ML, Phillips A, Shamir R, Troncone R, Giersiepen K, Branski D, Catassi C, Lelgeman M, Maki M, Ribes-Koninckx C, Ventura A, Zimmer KP; ESPGHAN Working Group on Coeliac Disease Diagnosis; ESPGHAN Gastroenterology Committee; European Society for Pediatric Gastroenterology, Hepatology, and Nutrition. European Society for Pediatric Gastroenterology, Hepatology, and Nutrition guidelines for the diagnosis of coeliac disease. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):136-60. doi: 10.1097/MPG.0b013e31821a23d0. PMID 22197856
- [Background] Bardella MT, Velio P, Cesana BM, Prampolini L, Casella G, Di Bella C, Lanzini A, Gambarotti M, Bassotti G, Villanacci V. Coeliac disease: a histological follow-up study. Histopathology. 2007 Mar;50(4):465-71. doi: 10.1111/j.1365-2559.2007.02621.x. PMID 17448022
- [Background] Holmes GK, Prior P, Lane MR, Pope D, Allan RN. Malignancy in coeliac disease--effect of a gluten free diet. Gut. 1989 Mar;30(3):333-8. doi: 10.1136/gut.30.3.333. PMID 2707633
- [Background] Kaukinen K, Peraaho M, Lindfors K, Partanen J, Woolley N, Pikkarainen P, Karvonen AL, Laasanen T, Sievanen H, Maki M, Collin P. Persistent small bowel mucosal villous atrophy without symptoms in coeliac disease. Aliment Pharmacol Ther. 2007 May 15;25(10):1237-45. doi: 10.1111/j.1365-2036.2007.03311.x. PMID 17451570
- [Background] Silano M, Volta U, Vincenzi AD, Dessi M, Vincenzi MD; Collaborating Centers of the Italian Registry of the Complications of Coeliac Disease. Effect of a gluten-free diet on the risk of enteropathy-associated T-cell lymphoma in celiac disease. Dig Dis Sci. 2008 Apr;53(4):972-6. doi: 10.1007/s10620-007-9952-8. Epub 2007 Oct 13. PMID 17934841
- [Background] Cosnes J, Cellier C, Viola S, Colombel JF, Michaud L, Sarles J, Hugot JP, Ginies JL, Dabadie A, Mouterde O, Allez M, Nion-Larmurier I; Groupe D'Etude et de Recherche Sur la Maladie Coeliaque. Incidence of autoimmune diseases in celiac disease: protective effect of the gluten-free diet. Clin Gastroenterol Hepatol. 2008 Jul;6(7):753-8. doi: 10.1016/j.cgh.2007.12.022. Epub 2008 Feb 6. PMID 18255352
- [Background] Castano L, Blarduni E, Ortiz L, Nunez J, Bilbao JR, Rica I, Martul P, Vitoria JC. Prospective population screening for celiac disease: high prevalence in the first 3 years of life. J Pediatr Gastroenterol Nutr. 2004 Jul;39(1):80-4. doi: 10.1097/00005176-200407000-00016. PMID 15187786
- [Background] Tanpowpong P, Broder-Fingert S, Katz AJ, Camargo CA Jr. Age-related patterns in clinical presentations and gluten-related issues among children and adolescents with celiac disease. Clin Transl Gastroenterol. 2012 Feb 16;3(2):e9. doi: 10.1038/ctg.2012.4. PMID 23238134
- [Background] Rubio-Tapia A, Hill ID, Kelly CP, Calderwood AH, Murray JA; American College of Gastroenterology. ACG clinical guidelines: diagnosis and management of celiac disease. Am J Gastroenterol. 2013 May;108(5):656-76; quiz 677. doi: 10.1038/ajg.2013.79. Epub 2013 Apr 23. PMID 23609613
- [Background] Dorn SD, Matchar DB. Cost-effectiveness analysis of strategies for diagnosing celiac disease. Dig Dis Sci. 2008 Mar;53(3):680-8. doi: 10.1007/s10620-007-9939-5. Epub 2007 Oct 13. PMID 17934849
- [Background] Collin P. Should adults be screened for celiac disease? What are the benefits and harms of screening? Gastroenterology. 2005 Apr;128(4 Suppl 1):S104-8. doi: 10.1053/j.gastro.2005.02.021. PMID 15825117
- [Background] Lagerqvist C, Dahlbom I, Hansson T, Jidell E, Juto P, Olcen P, Stenlund H, Hernell O, Ivarsson A. Antigliadin immunoglobulin A best in finding celiac disease in children younger than 18 months of age. J Pediatr Gastroenterol Nutr. 2008 Oct;47(4):428-35. doi: 10.1097/MPG.0b013e31817d80f4. PMID 18852634
- [Background] Korponay-Szabo IR, Dahlbom I, Laurila K, Koskinen S, Woolley N, Partanen J, Kovacs JB, Maki M, Hansson T. Elevation of IgG antibodies against tissue transglutaminase as a diagnostic tool for coeliac disease in selective IgA deficiency. Gut. 2003 Nov;52(11):1567-71. doi: 10.1136/gut.52.11.1567. PMID 14570724
- See also: Celiac Disease Early Diagnosis Protocol — https://www.mscbs.gob.es/profesionales/prestacionesSanitarias/publicaciones/Celiaquia/enfermedadCeliaca.pdf